CLINICAL TRIAL: NCT06338553
Title: Optimizing Stage 2 T1DM Management: Assessing the Impact of GLP-1Ra on Metabolic Outcomes in Patients Receiving Teplizumab
Brief Title: GLP-1Ra Impact on Metabolic Outcomes in Stage 2 T1DM While Receiving Teplizumab
Acronym: GLP-TEP
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Daniel Moore, Associate Professor of Pediatrics, Division of Pediatric Endocrinology and Diabetes, Vanderbilt University Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: 231620; R01DK139322 (NIH)
Record Dates: First submitted 2024-03-07; First posted 2024-03-29 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Type 1 Diabetes
Keywords: Type 1 Diabetes; Stage 2 Type 1 Diabetes; Early Stage Type 1 Diabetes; GLP1-Ra; Rybelsus; mixed meal tolerance test (MMTT); Stage 3 Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — semaglutide

STUDY DESIGN:
Intervention Model Description: In this study, participants with stage 2 T1DM undergoing Teplizumab treatment will be randomly assigned to receive single doses of either a GLP-1Ra (oral semaglutide, Rybelsus®) or a placebo, and three separate Mixed Meal Tolerance Test (MMTT) tests, 3-5 months apart, will be conducted to assess the effects on blood sugar levels, insulin function, and vascular health.
  Participants with early stage 3 T1DM will undergo four MMTT studies: two at baseline shortly after diagnosis and two after a six-month interval. During each pair of studies, participants will receive a single dose of GLP-1Ra (oral semaglutide, Rybelsus®) in one study and placebo in the other, with the order randomized to minimize potential sequencing effects. This approach allows us to assess the effects of GLP-1Ra on metabolic parameters and β-cell function at two critical time points in disease progression, shortly after diagnosis and after a six-month interval.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: For applicable participants, a placebo will be given prior to a pre-TZIELD® meal test. For participants who have already received Teplizumab (TZIELD®) or those who are progressing to the 2 remaining study visits, a GLP-1Ra or placebo will be given in random orders at these two visits. The GLP-1Ra will only be given one time.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- Participants receiving placebo, Stage 2 T1DM participants (Placebo Comparator): Participants receive a placebo orally once before the pre-TZIELD® MMTT. Participants also receive a placebo orally once before one of the post-TZIELD® MMTTs.
  Interventions: Drug: Placebo
- Participants receiving a semaglutide (Rybelsus®), Stage 2 T1DM participants (Experimental): Participants receive 7mg of semaglutide (Rybelsus®) orally once before one of the post-TZIELD® MMTTs. Rybelsus is only given one time.
  Interventions: Drug: Semaglutide (Rybelsus®)
- Placebo Comparator: Participants receiving placebo, Stage 3 T1DM participants (Placebo Comparator): Participants receive a placebo orally once before each MMTT.
  Interventions: Drug: Placebo
- Experimental: Participants receiving a semaglutide (Rybelsus®), Stage 3 T1DM participants (Experimental): Participants receive 7mg of semaglutide (Rybelsus®) orally once before each MMTT.
  Interventions: Drug: Semaglutide (Rybelsus®)

INTERVENTIONS:
Drug: Semaglutide (Rybelsus®) — 7 mg single dose of Rybelsus® by mouth once before each MMTT
  Arms: Experimental: Participants receiving a semaglutide (Rybelsus®), Stage 3 T1DM participants; Participants receiving a semaglutide (Rybelsus®), Stage 2 T1DM participants
Drug: Placebo — placebo capsule or tablet once before each MMTT.
  Arms: Participants receiving placebo, Stage 2 T1DM participants; Placebo Comparator: Participants receiving placebo, Stage 3 T1DM participants

SUMMARY:
The goal of this study is to determine how a drug class called glucagon-like peptide-1 receptor agonists (GLP-1Ra) affects people during an early stage of Type 1 Diabetes undergoing clinical teplizumab treatment. This study involves giving participants a liquid meal under different conditions and observing how their bodies respond, focusing on blood sugar levels, insulin effectiveness, and blood vessel function. The meal tests are followed by two post-treatment tests, one with the GLP-1Ra drug and the other with a placebo. Each test involves blood draws before and during the meal test, GLP-1Ra or placebo administration, and an ultrasound to measure blood vessel function. The goal is to see if GLP-1Ra can help manage blood sugar levels and improve cardiovascular health in this population.

DETAILED DESCRIPTION:
The long-term goal is to determine whether repurposing GLP-1Ra for stage 2 in combination with immunotherapy can modify the disease course, reducing the need for exogenous insulin therapy and leading to improved cardiometabolic outcomes and quality of life. For early stage 3 T1DM, we aim to determine whether GLP-1Ra can offer similar protective effects in preserving β-cell function and stabilizing glycemic control.

The immediate objective is to investigate the impact of GLP-1Ra's insulinotropic and glucagonostatic effects on dysmetabolism in stage 2 and early stage 3 T1DM. The study hypothesizes that these effects will each delay the need for exogenous insulin by improving three key aspects of dysmetabolism: 1) postprandial glycemia, 2) disposition index (i.e., the ability of the islet cells to compensate for a given insulin sensitivity), and 3) endothelial function. The rationale for this hypothesis is based on two observations: first, GLP-1Ra combined with immunomodulatory therapy sustains endogenous secretion in response to a mixed meal tolerance test (MMTT) during the first year of stage 3; and second, GLP-1Ras mitigate postprandial hyperglucagonemia in longer-duration T1DM. To test the hypothesis, studies will be conduct in individuals with stage 2 T1DM treated with teplizumab using a crossover design structured around the following specific aims:

Aim 1: Investigate the impact of GLP-1Ra on postprandial glycemia in a pilot study. The study team will measure postprandial glycemia during an MMTT before teplizumab treatment. After teplizumab the study team will compare the effects of placebo versus semaglutide (a GLP-1Ra).

Aim 2: Study the impact of GLP-1Ra on the disposition index (DI) in a pilot study. The study team will use the oral glucose minimal model to measure DI during an MMTT before and after teplizumab treatment, comparing the effects of placebo versus semaglutide. As an exploratory outcome, β-cell endoplasmic reticulum dysfunction will be quantified by measuring the proinsulin-to-C-peptide ratio during the MMTT.

Aim 3: Determine the impact of GLP-1Ra on endothelial function in a pilot study. The study team will use B-mode ultrasound to measure flow mediated vasodilation (FMD), a bioassay of endothelial function, during each MMTT. Because endothelial cells are often among the first affected by hyperglycemia and insulin resistance, the study aims to illuminate how GLP-1Ra may mitigate early vascular disease progression.

And in a pilot study of early stage 3 T1DM, 4) GLP-1 Receptor Agonists. Aim 4: Determine how much GLP-1Ra monotherapy therapy changes the disposition index (DI) in a pilot study of early stage 3 T1DM.

Despite the promise of TZIELD®, the medication is not currently approved for patients with stage 3 T1DM. Thus, individuals who progress into stage 3 T1DM continue to face significant challenges, including loss of β-cell function and the need for exogenous insulin. As patients move into stage 3, there is an opportunity for metabolic interventions that may preserve residual insulin production and mitigate the long-term impact of hyperglycemia. Accordingly, we will conduct a randomized, double-blind, placebo-controlled crossover study involving patients with early stage 3 T1DM. Each participant will undergo four mixed meal tolerance tests (MMTTs): two at baseline shortly after diagnosis and two after a six-month interval. During each MMTT, participants will receive either a single dose of GLP-1Ra (oral semaglutide) or placebo in a randomized order. This design allows us to assess the independent effects of GLP-1Ra on the disposition index (DI) by comparing the results between the GLP-1Ra and placebo conditions at both time points. By evaluating changes in DI and other metabolic parameters over time, we aim to determine how GLP-1Ra monotherapy influences β-cell function and insulin sensitivity in early stage 3 T1DM.

ELIGIBILITY:
Aims 1-3: Stage 2 T1DM with TZIELD® and GLP-1Ra

Inclusion Criteria:

* Age: 12-50 years
* BMI: 18-31 kg/m2 (adults) or 5-95th %ile (pediatric)
* Stage 2 T1DM (i.e., ≥ 2 islet auto-antibodies and:
* fasting glucose ≥ 100 mg/dL and < 126 mg/dL OR
* 2-hr OGTT /MMTT ≥ 140 mg/dL and < 200 mg/dL OR
* During an OGTT having a glucose of > 199 mg/dL at 30, 60, or 90 minutes)

Exclusion Criteria:

* Comorbidities:
* SBP > 140 mmHg and DBP > 100 mmHg
* eGFR by MDRD equation of < 60 mL/min/1.73m2
* AST or ALT > 2.5 times ULN
* Family history of medullary thyroid carcinoma
* Diagnosis of pancreatitis or gastroparesis within the past 3 years
* Medications: Any diabetes medication, any antioxidant vitamin supplement (<2 weeks before a study), any systemic glucocorticoid, antipsychotic, atenolol, metoprolol, propranolol, niacin, any thiazide diuretic, any OCP with > 35 mcg ethinyl estradiol, growth hormone, any immunosuppressant, antihypertensive, any antihyperlipidemic
* Other: pregnancy, peri- or post-menopausal women, active smoker

Aim 4: Early Stage 3 T1DM with GLP-1Ra Monotherapy Inclusion Criteria

* Age: 12-50 years
* BMI: 18-31 kg/m2 (adults) or 5-95th %ile (pediatric)
* Early stage 3 T1DM with either
* HbA1c 6.5% to 8.0% at diagnosis OR
* HbA1c 5.7% to 6.4% with oral glucose test meeting ADA criteria for stage 3 T1DM within the past three months prior to or during screening visit
* Time of stage 3 diagnosis: within eight weeks of first study visit

Exclusion Criteria

* DKA history: history of diabetic ketoacidosis requiring hospital admission
* Comorbidities:
* Family history of medullary thyroid carcinoma
* Diagnosis of pancreatitis or gastroparesis within the past 3 years
* Medications: Any diabetes medication, any antioxidant vitamin supplement (<2 weeks before a study), any systemic glucocorticoid, antipsychotic, atenolol, metoprolol, propranolol, niacin, any thiazide diuretic, any OCP with > 35 mcg ethinyl estradiol, growth hormone, any immunosuppressant, antihypertensive, any antihyperlipidemic
* Other: pregnancy, peri- or post-menopausal women, active smoker

Ages: 12 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Investigate the impact of GLP-1Ra on postprandial glycemia in a pilot study | During the MMTT in which the participant is randomly selected to receive semaglutide (Rybelsus®), glucose level will be checked at timepoints -30, -15, 0, 10, 20, 30, 60, 90, 120, 150, 180, and 240 minutes
  Researchers will measure postprandial glycemia during an MMTT before TZIELD® treatment. After TZIELD®, the effects of placebo versus semaglutide (Rybelsus®),a GLP-1Ra, will be compared.
Study the impact of GLP-1Ra on the disposition index (DI) in a pilot study | Based on the glucose and insulin readings obtained at timepoints -30, -15, 0, 10, 20, 30, 60, 90, 120, 150, 180, and 240 min and calculated approximately 1 month following completion of the MMTT once insulin levels in plasma are resulted.
  Researchers will use the oral glucose minimal model to measure DI during an MMTT before and after TZIELD® treatment, comparing the effects of placebo versus Rybelsus®. As an exploratory outcome, β-cell endoplasmic reticulum dysfunction will be determined by measuring the proinsulin-to-C-peptide ratio during the MMTT.
Determine the impact of GLP-1Ra on endothelial function in a pilot study | During the last 30 minutes of each MMTT, between the 210 and 240 timepoints
  B-mode ultrasound will be used to measure flow-mediated vasodilation (FMD), a bioassay of endothelial function, during each MMTT. Because endothelial cells are often among the first affected by hyperglycemia and insulin resistance, researchers aim to illuminate how GLP-1Ra may mitigate early vascular disease progression.
Determine how much GLP-1Ra monotherapy therapy changes the disposition index (DI) in a pilot study of early stage 3 T1DM. | During the MMTT in which the participant is randomly selected to receive semaglutide (Rybelsus®), glucose level will be checked at timepoints -30, -15, 0, 10, 20, 30, 60, 90, 120, 150, 180, and 240 minutes
  Researchers will assess the independent effects of GLP-1Ra on the disposition index (DI) by comparing the results between the GLP-1Ra and placebo conditions during four mixed meal tolerance tests (MMTTs): two at baseline shortly after diagnosis and two after a six-month interval.

CONTACTS AND LOCATIONS:
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this study may be provided to qualified researchers with academic interest in type 1 diabetes. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, ICF
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis.
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA).

DOCUMENTS (1):
  • Study Protocol (2025-10-23): https://cdn.clinicaltrials.gov/large-docs/53/NCT06338553/Prot_004.pdf